CLINICAL TRIAL: NCT04364269
Title: A Phase 2a, Double-blind, Randomised, Placebo-controlled, Parallel Group, Multicentre Study on Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Multiple Doses of VIT-2763 in Subjects With Non-transfusion Dependent β-thalassaemia
Brief Title: Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) and Preliminary Efficacy of VIT-2763 in β-thalassaemia
Acronym: VITHAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vifor (International) Inc. (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIT-2763-THAL-201; 2019-002221-29 (EudraCT Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-28 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Beta-Thalassemia; Non-transfusion-dependent Thalassemia
Keywords: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — BID protein, human

STUDY DESIGN:
Intervention Model Description: Multiple dose, multicenter, double-blind, placebo-controlled parallel group study in adult and adolescent male and female subjects with non-transfusion dependent thalassemia (NTDT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will receive a randomisation number using a validated centralised procedure (IWRS) that automates the random assignment of treatment groups to randomisation numbers. The randomisation plan will be kept strictly confidential, accessible only to authorised persons, until the time of unblinding.
  The study drugs (VIT-2763 or placebo) are provided in identical white opaque hard capsules in packaging of identical appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VIT-2763 Once a day (QD) (Experimental): Participants will be assigned to receive VIT-2763 once a day (QD) in a total daily dose of 60 mg or 120 mg depending on their body weight.
  The study medication (VIT-2763 and/or matching placebo) will be administered for all participants twice a day to maintain the blind.
  Interventions: Drug: VIT-2763 once a day (QD)
- VIT-2763 Twice a day (BID) (Experimental): Participants will be assigned to receive VIT-2763 Twice a day (BID) in a total daily dose of 60 mg or 120 mg depending on their body weight.
  Interventions: Drug: VIT-2763 twice a day (BID)
- Placebo (Placebo Comparator): Participants will be assigned to receive Placebo, Twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIT-2763 once a day (QD) — Participants will receive VIT-2763 QD at a dose of 60 mg if their body weight is between 40 kg to 59 kg or at a dose of 120 mg if their body weight is between 60 kg and 100 kg, during 12 weeks.
  Arms: VIT-2763 Once a day (QD)
Drug: VIT-2763 twice a day (BID) — Participants will receive VIT-2763 BID at a dose of 60 mg if their body weight is between 40 kg to 59 kg or at a dose of 120 mg if their body weight is between 60 kg and 100 kg, during 12 weeks.
  Arms: VIT-2763 Twice a day (BID)
Drug: Placebo — Participants will receive hard capsules of Placebo, twice a day.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled parallel group trial to investigate the safety, tolerability and efficacy of multiple doses of VIT-2763 versus placebo in participants with non-transfusion-dependent Beta-thalassemia (NTDT).

DETAILED DESCRIPTION:
The study includes a 12-week treatment period and a safety follow-up period of 4 weeks.

About 36 participants (adults and adolescents) are expected to take part in this study at a number of different institutions internationally.

Adult Participants (Cohort I) will be randomized to receive either VIT-2763 once daily (QD) or twice daily (BID) or placebo, at a dose of 120 mg or 60mg depending on their body weight. Following cohort I review, adolescent participants (Cohort II) will be randomized to the same study arms with the same interventions.

The study medication will be given as oral capsules, containing 60 mg of VIT-2763 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of NTDT, including a β-thalassemia intermedia-phenotype.
* NTDT is defined as subjects having received less than 5 units of red blood cells (RBCs) during the 24-week period prior to randomisation/first drug administration of VIT-2763 or placebo (Day 1; 1 unit is defined as 200 to 350 ml of transfused packed RBCs and last RBC transfusion must have been received at east 14 days prior to randomisation).
* Male and female adult NTDT subjects, 18-65 years of age inclusive (Cohort I only) at time of screening.
* Male and female adolescent NTDT subjects, 12-17 years of age inclusive (Cohort II only) at time of screening.
* Subjects must have a mean baseline hemoglobin (Hb) equal to or lower than 11 g/dl, based on at least 2 consecutive measurements with at least 1 week apart within 6 weeks prior to randomisation/baseline.

Exclusion Criteria:

* Documented diagnosis of transfusion dependent thalassemia (TDT), including a beta-thalassemia major phenotype (including β0/β0, β+/β+, β0/β+ genotype), and mixed compound heterozygous for sickling phenotype variants such as Hb S/β- thalassemia, or transfusion dependent non-deletional Hb H disease (i.e., Hb constant spring) or Hb C disease.
* Subjects on concomitant iron chelation therapy (ICT) or subjects on prior ICT when discontinued less than 4 weeks prior randomisation. If ICT was discontinued at least 4 weeks prior randomization the subject is eligible.
* ICT naïve subjects or subjects who discontinued ICT therapy at least 6 months before the screening visit with serum ferritin lower than 150 ng/ml and/or documented liver iron concentration (LIC) equal to or lower than 1 mg/g liver dry weight assessed through magnetic resonance imaging (MRI), or subjects on prior ICT with serum ferritin lower than 300 ng/ml and/or documented LIC lower than 3 mg/g liver dry weight assessed through MRI.
* Subjects with transferrin saturation (TSAT) less than 30%.
* Subjects with documented LIC greater than 15 mg/g liver dry weight assessed through MRI, or a documented myocardial T2* less than 20 ms, if available per local practice and retrieved within 24 months prior to randomization.
* Adult or adolescent subjects with body weight lower than 40.0 kg or greater than 100 kg at screening.
* Chronic liver disease and/or alanine transaminase (ALT), aspartate transaminase (AST) or gamma-glutamyl transpeptidase (GGT) above 3-fold the upper limit of normal (ULN) range at screening.
* Estimated glomerular filtration rate (eGFR) less than 30 ml/min/1.73 m2 (according to chronic kidney disease classification Stage 4 or higher), and/or significant albuminuria greater than 30 mg/mmol. eGFR should be estimated according to Chronic Kidney Disease Epidemiology Collaboration formula (CKI-EPI) in adults, and Schwartz formula in adolescents.
* Newly diagnosed folate deficiency anemia and/or Vitamin B12 megaloblastic anemia. Subjects with known folate deficiency anemia and/or Vitamin B12 megaloblastic anemia who are on at least 12 weeks stable replacement therapy are eligible.
* Any history or clinically important finding of cardiac disorders, such as clinically relevant cardiac arrhythmia, cardiomyopathy, coronary disease, valve disorder, or heart failure according to New York Heart Association classification 3-4.
* Subjects with history of partial or total splenectomy within 6 months prior to screening.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Department, Study Director — Vifor (International) Inc.
Locations (16):
- Greece (3):
  - Clinical Site #301, Athens, Attica
  - Clinical Site #302, Rio
  - Clinical Site #303, Thessaloniki
- Israel (3):
  - Clinical Site #401, Afula
  - Clinical Site #402, Haifa
  - Clinical Site #403, Petah Tikva
- Italy (6):
  - Clinical Site #201, Milan, MI
  - Clinical Site #203, Napoli
  - Clinical Site #206, Napoli
  - Clinical Site #207, Orbassano
  - Clinical Site #205, Palermo
  - Clinical Site #202, Verona
- Clinical Site #101, Beirut, Lebanon
- Thailand (3):
  - Clinical Site #501, Bangkok
  - Clinical Site #502, Chiang Mai
  - Clinical Site #503, Phitsanulok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kattamis A, Taher A, Viprakasit V, Levin C, Hermosilla R, Szecsody P, Richard F, Cappellini MD, Porter J. Safety and pharmacodynamics of the ferroportin inhibitor vamifeport in patients with non-transfusion-dependent beta-thalassemia: results from a randomized phase 2a study. Orphanet J Rare Dis. 2025 Nov 25;20(1):608. doi: 10.1186/s13023-025-04119-y. PMID 41291806

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From a total of 35 screened participants, 25 were randomized in the study. A total of 10 participants were not randomised, among which 2 participants withdrew their consent, and 8 participants did not meet the inclusion criteria.
Groups:
- VIT-2763 QD: Participants who received VIT-2763 once a day (QD) in a total daily dose of 60 mg or 120 mg, depending on their body weight, during 12 weeks.
  Participants received VIT-2763 QD at a dose of 60 mg if their body weight was between 40 kg to 59 kg or at a dose of 120 mg if their body weight was between 60 kg and 100 kg.
  The study medication (VIT-2763 and/or matching placebo) was administered to all participants twice a day to maintain the blind.
  QD = once a day
- VIT-2763 BID: Participants who received VIT-2763 twice a day (BID) in a total daily dose of 60 mg or 120 mg, depending on their body weight, during 12 weeks.
  Participants received VIT-2763 BID at a dose of 60 mg if their body weight was between 40 kg to 59 kg or at a dose of 120 mg if their body weight was between 60 kg and 100 kg.
  BID = twice a day
- Placebo: Participants who received twice a day hard capsules of placebo, during 12 weeks.
Period: Overall Study
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Started | 9 | 12 | 4
Completed | 8 | 11 | 4
Not Completed | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo | Total
Number analyzed (Participants) | 9 | 12 | 4 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 4 | 25
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 1 | 9
  Male | 3 | 10 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 11 | 4 | 24
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 3 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 9 | 3 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 3 | 3 | 1 | 7
  Lebanon | 1 | 2 | 0 | 3
  Italy | 0 | 3 | 0 | 3
  Israel | 0 | 1 | 2 | 3
  Thailand | 5 | 3 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Please note that in this section we are presenting just the overview of the adverse events experienced by the trial participants, in particular, the number of participants with at least one TEAE. Please refer to the detailed tables included on the Adverse Event Module for specifics.
Time Frame: From baseline to Week 16
Population: The safety set (SS) was defined as all randomized participants who had taken at least 1 dose of study medication. The participants in the SS were to be analyzed based on the treatment they received, regardless of randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
Participants | 6 | 7 | 3

2. Primary Outcome: Changes in the Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Summary of the values by visit from baseline and changes from baseline by post-baseline visit.
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
millimeters of mercury (mmHg)
  SBP Baseline | 114.2 (11.62) | 114.7 (13.88) | 114.8 (12.97)
  SBP Week 1 | 115.0 (8.35) | 116.7 (10.65) | 104.0 (8.98)
  SBP Change from Baseline to Week 1 | 0.8 (8.94) | 2.0 (9.72) | -10.8 (10.90)
  SBP Week 2 | 113.9 (9.41) | 118.3 (14.85) | 114.8 (15.06)
  SBP Change from Baseline to Week 2 | -0.3 (6.60) | 3.6 (8.78) | 0.0 (2.83)
  SBP Week 4 | 112.0 (11.20) | 113.9 (12.41) | 104.8 (6.85)
  SBP Change from Baseline to Week 4 | -2.2 (8.77) | -0.8 (8.51) | -10.0 (14.72)
  SBP Week 8 | 114.9 (7.41) | 113.8 (10.54) | 109.8 (12.61)
  SBP Change from Baseline to Week 8 | 0.7 (11.11) | 0.9 (9.63) | -5.0 (1.63)
  SBP Week 12 | 113.4 (11.02) | 112.8 (11.31) | 107.5 (10.08)
  SBP Change from Baseline to Week 12 | -0.8 (13.02) | -0.1 (10.85) | -7.3 (3.40)
  DBP Baseline | 65.94 (10.088) | 65.00 (10.189) | 66.50 (7.853)
  DBP Week 1 | 66.44 (6.710) | 69.33 (9.921) | 61.75 (4.856)
  DBP Change from Baseline to Week 1 | 0.50 (4.886) | 4.33 (6.344) | -4.75 (6.185)
  DBP Week 2 | 65.89 (9.545) | 68.83 (11.535) | 64.00 (6.055)
  DBP Change from Baseline to Week 2 | -0.06 (5.353) | 3.83 (8.726) | -2.50 (3.000)
  DBP Week 4 | 65.22 (11.043) | 62.33 (9.069) | 62.75 (3.775)
  DBP Change from Baseline to Week 4 | -0.72 (9.398) | -2.67 (9.921) | -3.75 (5.058)
  DBP Week 8 | 63.44 (6.579) | 67.18 (9.174) | 66.75 (7.500)
  DBP Change from Baseline to Week 8 | -2.50 (8.216) | 3.27 (8.439) | 0.25 (7.848)
  DBP Week 12 | 63.67 (7.697) | 67.64 (9.657) | 62.50 (3.317)
  DBP Change from Baseline to Week 12 | -2.28 (10.140) | 3.73 (6.310) | -4.00 (6.880)

3. Primary Outcome: Changes in the Heart Rate
Description: Summary of the values by visit from baseline and changes from baseline by post-baseline visit.
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Pulse Rate (bpm)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
Pulse Rate (bpm)
  Baseline | 82.00 (12.135) | 77.71 (10.208) | 73.75 (5.560)
  Week 1 | 82.33 (11.694) | 80.33 (9.875) | 70.75 (6.449)
  Change from Baseline to Week 1 | 0.33 (6.042) | 2.63 (5.859) | -3.00 (5.715)
  Week 2 | 83.56 (12.856) | 75.83 (9.953) | 75.00 (8.756)
  Change from Baseline to Week 2 | 1.56 (10.442) | -1.88 (8.263) | 1.25 (3.775)
  Week 4 | 82.33 (14.414) | 77.92 (9.830) | 73.25 (3.775)
  Change from Baseline to Week 4 | 0.33 (8.818) | 0.21 (5.541) | -0.50 (1.915)
  Week 8 | 83.22 (11.322) | 80.27 (10.992) | 72.50 (5.196)
  Change from Baseline to Week 8 | 1.22 (6.648) | 2.68 (9.040) | -1.25 (7.411)
  Week 12 | 81.44 (9.002) | 79.91 (8.734) | 74.25 (4.193)
  Change from Baseline to Week 12 | -0.56 (8.719) | 2.32 (9.419) | 0.50 (6.137)

4. Primary Outcome: Changes in 12-lead Electrocardiogram (ECG) Parameters
Description: Values by visit from baseline and changes from baseline by post-baseline visit. The following ECG parameters were recorded: PR interval, QRS duration, QT interval, RR interval and QTcF interval.
  PR interval represents the time from the onset of the P wave to the start of the QRS complex. QRS duration represents the time required for a stimulus to spread through the ventricles (ventricular depolarization). QT interval represents the time from the start of the Q wave to the end of the T wave. RR interval represents the time from the onset of one R wave to the onset of the next one, one complete cardiac cycle. QT corrected for heart rate (QTc) interval reflects ventricular repolarization.
Time Frame: From baseline to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
milliseconds (ms)
  PR interval - Baseline | 158.3 (25.14) | 147.6 (20.05) | 175.8 (38.92)
  PR interval - Baseline 2h post-dose | 161.2 (21.28) | 155.1 (17.98) | 175.0 (14.07)
  PR interval - Change from Baseline to Baseline 2h post-dose | 2.9 (25.78) | 6.3 (16.45) | -0.8 (38.59)
  PR interval - Week 1 | 159.2 (22.90) | 153.0 (14.12) | 189.5 (18.72)
  PR interval - Change from Baseline to Week 1 | 0.9 (16.59) | 4.7 (12.71) | 13.8 (25.67)
  PR interval - Week 2 | 167.6 (26.49) | 153.0 (17.87) | 185.5 (4.43)
  PR interval - Change from Baseline to Week 2 | 9.2 (27.64) | 5.5 (13.56) | 9.8 (37.56)
  PR interval - Week 4 | 154.0 (26.49) | 154.2 (21.19) | 185.0 (7.39)
  PR interval - Change from Baseline to Week 4 | -4.3 (18.85) | 8.1 (15.48) | 9.3 (33.42)
  PR interval - Week 8 | 161.2 (19.34) | 153.5 (20.61) | 185.8 (10.14)
  PR interval - Change from Baseline to Week 8 | 2.9 (17.05) | 7.1 (12.66) | 10.0 (32.86)
  PR interval - Week 12 | 160.6 (19.55) | 156.6 (14.47) | 182.8 (11.98)
  PR interval - Change from Baseline to Week 12 | 2.2 (19.50) | 11.5 (14.25) | 7.0 (36.09)
  QRS duration - Baseline | 94.0 (18.73) | 88.8 (19.17) | 119.3 (50.12)
  QRS duration - Baseline 2h post-dose | 94.3 (20.21) | 95.8 (10.96) | 85.0 (11.60)
  QRS duration - Change from Baseline to Baseline 2h post-dose | 0.3 (4.82) | 7.0 (14.39) | -34.3 (55.27)
  QRS duration - Week 1 | 98.4 (23.16) | 96.1 (11.27) | 98.0 (16.57)
  QRS duration - Change from Baseline to Week 1 | 4.4 (14.75) | 7.3 (13.45) | -21.3 (65.76)
  QRS duration - Week 2 | 94.0 (29.01) | 96.3 (14.13) | 91.3 (12.09)
  QRS duration - Change from Baseline to Week 2 | 0.0 (23.04) | 7.6 (17.96) | -28.0 (61.36)
  QRS duration - Week 4 | 92.3 (23.32) | 92.6 (15.11) | 94.3 (8.10)
  QRS duration - Change from Baseline to Week 4 | -1.7 (11.16) | 6.0 (16.76) | -25.0 (54.02)
  QRS duration - Week 8 | 91.0 (24.72) | 94.9 (18.27) | 93.3 (10.81)
  QRS duration - Change from Baseline to Week 8 | -3.0 (15.99) | 7.4 (28.52) | -26.0 (60.02)
  QRS duration - Week 12 | 94.3 (27.31) | 84.8 (18.66) | 91.8 (10.59)
  QRS duration - Change from Baseline to Week 12 | 0.3 (20.64) | -2.7 (23.70) | -27.5 (60.69)
  QT interval - Baseline | 371.7 (76.41) | 374.2 (21.78) | 420.8 (48.75)
  QT interval - Baseline 2h post-dose | 385.7 (50.89) | 376.8 (22.25) | 379.5 (30.17)
  QT interval - Change from Baseline to Baseline 2h post-dose | 14.0 (61.00) | 2.6 (21.49) | -41.3 (68.30)
  QT interval - Week 1 | 394.1 (47.36) | 374.8 (33.12) | 381.5 (32.18)
  QT interval - Change from Baseline to Week 1 | 22.4 (57.20) | 0.7 (28.96) | -39.3 (71.63)
  QT interval - Week 2 | 384.0 (55.52) | 367.0 (24.68) | 378.3 (27.89)
  QT interval - Change from Baseline to Week 2 | 12.3 (76.14) | -7.2 (27.61) | -42.5 (61.87)
  QT interval - Week 4 | 370.1 (67.13) | 373.6 (21.22) | 378.0 (36.51)
  QT interval - Change from Baseline to Week 4 | -1.6 (23.07) | 0.9 (24.94) | -42.8 (61.50)
  QT interval - Week 8 | 389.7 (39.20) | 379.4 (25.08) | 381.8 (37.99)
  QT interval - Change from Baseline to Week 8 | 18.0 (69.60) | 4.6 (22.59) | -39.0 (64.59)
  QT interval - Week 12 | 380.9 (59.97) | 364.2 (36.22) | 388.3 (42.85)
  QT interval - Change from Baseline to Week 12 | 9.2 (33.53) | -10.5 (33.69) | -32.5 (72.06)
  RR interval - Baseline | 789.4 (128.89) | 801.4 (95.56) | 877.5 (114.65)
  RR interval - Baseline 2h post-dose | 781.2 (155.21) | 805.5 (119.36) | 812.5 (124.38)
  RR interval - Change from Baseline to Baseline 2h post-dose | -8.2 (87.78) | 4.1 (112.91) | -65.0 (196.09)
  RR interval - Week 1 | 793.2 (105.35) | 864.9 (149.33) | 826.5 (96.57)
  RR interval - Change from Baseline to Week 1 | 3.8 (82.82) | 63.5 (137.59) | -51.0 (98.80)
  RR interval - Week 2 | 757.3 (120.25) | 830.1 (138.34) | 833.8 (16.01)
  RR interval - Change from Baseline to Week 2 | -32.1 (146.70) | 28.7 (117.34) | -43.8 (103.92)
  RR interval - Week 4 | 783.7 (110.55) | 829.8 (154.72) | 825.8 (96.08)
  RR interval - Change from Baseline to Week 4 | -5.8 (62.11) | 34.1 (137.64) | -51.8 (111.05)
  RR interval - Week 8 | 765.0 (91.52) | 810.1 (138.16) | 844.8 (135.47)
  RR interval - Change from Baseline to Week 8 | -24.4 (116.42) | 17.2 (108.39) | -32.8 (152.45)
  RR interval - Week 12 | 780.7 (140.88) | 812.9 (93.89) | 878.3 (133.70)
  RR interval - Change from Baseline to Week 12 | -8.8 (115.95) | 20.0 (73.46) | 0.8 (172.81)
  QTcF interval - Baseline | 403.3 (80.48) | 400.5 (22.76) | 416.8 (17.46)
  QTcF interval - Baseline 2h post-dose | 419.3 (36.58) | 410.1 (25.34) | 407.3 (13.05)
  QTcF interval - Change from Baseline to Baseline 2h post-dose | 16.0 (66.51) | 9.6 (22.60) | -9.5 (6.76)
  QTcF interval - Week 1 | 425.7 (37.25) | 397.3 (30.44) | 406.8 (26.02)
  QTcF interval - Change from Baseline to Week 1 | 22.3 (65.53) | -3.3 (24.92) | -10.0 (20.38)
  QTcF interval - Week 2 | 420.8 (42.28) | 393.3 (28.90) | 402.0 (30.30)
  QTcF interval - Change from Baseline to Week 2 | 17.4 (77.84) | -7.2 (27.52) | -14.8 (14.52)
  QTcF interval - Week 4 | 401.3 (64.21) | 401.8 (27.41) | 402.8 (23.63)
  QTcF interval - Change from Baseline to Week 4 | -2.0 (24.74) | 2.1 (24.41) | -14.0 (7.07)
  QTcF interval - Week 8 | 426.0 (30.12) | 399.6 (27.17) | 404.3 (19.86)
  QTcF interval - Change from Baseline to Week 8 | 22.7 (80.36) | 0.3 (26.86) | -12.5 (4.51)
  QTcF interval - Week 12 | 414.1 (53.40) | 391.4 (42.91) | 405.3 (25.71)
  QTcF interval - Change from Baseline to Week 12 | 10.8 (37.94) | -8.0 (37.96) | -11.5 (10.63)

5. Secondary Outcome: Change From Baseline in Total Serum Iron
Description: Assessment of total serum Iron from baseline over a 12-week period (absolute and change from baseline).
  For the serum iron parameter, the 'Baseline' was collected during the screening period within the biochemistry sample.
Time Frame: From baseline to Week 12
Population: The full analysis set (FAS) was defined as all participants who were randomized to treatment, received at least one dose of randomized treatment and had at least one post-baseline pharmacodynamic assessment. The FAS was created in accordance with the intent-to-treat principles. The participants in the FAS were to be analyzed based on the treatment that they were randomized to.
Measure: Mean (Standard Deviation); unit: Micromoles per Litre (umol/L)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
Micromoles per Litre (umol/L)
  Baseline | 23.81 (13.438) | 28.42 (9.796) | 30.88 (13.329)
  Week 1 | 12.54 (9.159) | 11.38 (7.693) | 28.20 (17.919)
  Change from Baselines to Week 1 | -11.27 (7.158) | -17.03 (9.611) | -2.68 (12.365)
  Week 2 | 11.71 (8.622) | 12.99 (8.978) | 32.48 (15.541)
  Change from Baseline to Week 2 | -9.74 (4.707) | -15.43 (12.784) | 1.60 (3.996)
  Week 4 | 13.90 (12.222) | 12.85 (7.583) | 31.08 (13.721)
  Change from Baseline to Week 4 | -9.33 (4.659) | -14.03 (8.432) | 0.20 (2.902)
  Week 8 | 11.35 (7.822) | 11.55 (9.651) | 26.70 (12.040)
  Change from Baseline to Week 8 | -11.88 (9.627) | -17.05 (11.936) | -0.37 (3.550)
  Week 12 | 13.72 (11.031) | 11.62 (6.442) | 27.10 (12.856)
  Change from Baseline to Week 12 | -10.54 (6.782) | -16.22 (10.892) | 0.03 (2.701)

6. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Assessment of serum ferritin from baseline over a 12-week period (absolute and change from baseline).
  For the serum ferritin parameter, the 'Baseline' was collected during the screening period within the biochemistry sample.
Time Frame: From baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Microgrammes per Litre (ug/L)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
Microgrammes per Litre (ug/L)
  Baseline | 403.14 (226.315) | 1133.23 (2119.115) | 440.03 (321.453)
  Week 1 | 416.76 (220.567) | 471.53 (209.800) | 445.80 (228.244)
  Change from Baseline to Week 1 | -10.14 (31.509) | 40.89 (164.466) | 5.77 (93.946)
  Week 2 | 441.34 (269.599) | 500.79 (230.076) | 411.35 (207.477)
  Change from Baseline to Week 2 | 3.29 (60.579) | 23.80 (149.147) | -49.80 (76.867)
  Week 4 | 476.60 (282.457) | 585.71 (311.224) | 389.83 (240.553)
  Change from Baseline to Week 4 | 1.05 (61.638) | 89.98 (249.397) | -50.20 (80.958)
  Week 8 | 463.67 (206.646) | 508.56 (211.366) | 340.23 (165.356)
  Change from Baseline to Week 8 | -11.88 (43.063) | 52.84 (157.952) | -9.45 (20.577)
  Week 12 | 465.72 (227.378) | 927.42 (1478.471) | 261.70 (53.033)
  Change from Baseline to Week 12 | -15.84 (66.208) | -139.23 (626.380) | 7.25 (57.205)

7. Secondary Outcome: Change From Baseline in Serum Transferrin
Description: Assessment of serum transferrin from baseline over a 12-week period (absolute and change from baseline).
  For the serum transferrin parameter, the "Baseline 2h post-dose" was defined as the value at Visit 3 2h post-dose.
Time Frame: From baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Grammes per Litre (g/L)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
Grammes per Litre (g/L)
  Baseline 2h post-dose | 1.601 (0.4377) | 1.673 (0.3177) | 1.655 (0.3003)
  Week 1 | 1.610 (0.4557) | 1.822 (0.3903) | 1.683 (0.2210)
  Change from Baseline to Week 1 | 0.009 (0.1184) | 0.149 (0.1334) | 0.028 (0.2419)
  Week 2 | 1.601 (0.5043) | 1.759 (0.3569) | 1.655 (0.2408)
  Change from Baseline to Week 2 | -0.014 (0.1516) | 0.087 (0.1429) | 0.000 (0.1846)
  Week 4 | 1.708 (0.2672) | 1.705 (0.3496) | 1.745 (0.3756)
  Change from Baseline to Week 4 | 0.053 (0.2014) | 0.054 (0.1535) | 0.090 (0.2740)
  Week 8 | 1.640 (0.2745) | 1.725 (0.3194) | 1.553 (0.2836)
  Change from Baseline to Week 8 | -0.015 (0.0675) | 0.093 (0.1618) | -0.120 (0.0854)
  Week 12 | 1.706 (0.1954) | 1.656 (0.2974) | 1.610 (0.4784)
  Change from Baseline to Week 12 | -0.040 (0.1116) | 0.100 (0.1044) | -0.063 (0.1266)

8. Secondary Outcome: Change From Baseline in Calculated Transferrin Saturation (TSAT) )
Description: Assessment of TSAT from baseline over a 12-week period (absolute and change from baseline).
  For the calculated transferrin saturation parameter, the 'Baseline' was collected during the screening period within the biochemistry sample.
  Transferrin Saturation (TSAT) was calculated as Total Iron /Total Iron Binding Capacity (TIBC) X 100.
Time Frame: From baseline to Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: TSAT Percentage (%)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
Number analyzed (Participants) | 9 | 12 | 4
TSAT Percentage (%)
  Baseline | 69.3 (31.16) | 79.0 (24.05) | 83.3 (33.50)
  Week 1 | 36.8 (24.44) | 32.2 (21.44) | 56.5 (30.56)
  Change from Baselone to Week 1 | -32.6 (19.55) | -46.8 (22.55) | -26.8 (28.77)
  Week 2 | 36.0 (22.81) | 35.8 (24.13) | 71.5 (33.91)
  Change from Baseline to Week 2 | -29.5 (14.57) | -43.2 (33.23) | -11.8 (23.50)
  Week 4 | 41.0 (32.27) | 38.4 (24.85) | 82.5 (35.00)
  Change from Baseline to Week 4 | -24.0 (18.21) | -38.7 (27.57) | -0.8 (1.50)
  Week 8 | 32.3 (17.48) | 33.5 (27.08) | 77.3 (39.26)
  Change from Baseline to Week 8 | -32.7 (25.80) | -47.9 (29.70) | -0.3 (0.58)
  Week 12 | 36.0 (25.93) | 34.8 (17.76) | 76.3 (40.99)
  Change from Baseline to Week 12 | -27.6 (20.37) | -46.8 (23.61) | -1.3 (2.31)

9. Secondary Outcome: Pharmacokinetics Parameters - VIT-2763 Plasma Concentration Over Time
Description: Sparse sampling for determination of VIT-2763 plasma concentration following multiple dosing was obtained from pre-dose trough to 3 hours or 4 hours post-dose at selected study visits. Pharmacokinetics parameters (Cmax, clearance, distribution volume, area under the curve (AUC) were not calculated for the study.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | VIT-2763 QD | VIT-2763 BID
Number analyzed (Participants) | 9 | 12
nanograms per milliliter (ng/mL)
  Visit 3 1 hour post-dose | 796.5 (508.2) | 609.6 (455.2)
  Visit 3 4 hours post-dose | 222.3 (73.1) | 411.0 (269.5)
  Visit 6 pre-dose | 17.2 (10.2) | 114.4 (78.2)
  Visit 6 1 hour post-dose | 986.2 (796.7) | 483.5 (247.3)
  Visit 6 3 hours post-dose | 578.2 (494.5) | 544.3 (337.5)
  Visit 7 pre-dose | 15.5 (6.6) | 111.0 (61.9)
  Visit 7 1 hour post-dose | 751.7 (682.3) | 692.2 (470.2)
  Visit 7 4 hours post-dose | 295.5 (209.5) | 384.3 (200.9)
  Visit 8 pre-dose | 361.5 (579.2) | 136.0 (76.8)
  Visit 8 1 hour post-dose | 894.1 (670.3) | 650.6 (474.5)
  Visit 8 3 hours post-dose | 684.0 (405.5) | 569.9 (343.1)

ADVERSE EVENTS:
Time Frame: up to 20 weeks (all visits/phone calls through study completion are considered)
Arm/Group | VIT-2763 QD | VIT-2763 BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/4
Other Adverse Events (participants affected / at risk) | 6/9 | 7/12 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIT-2763 QD (N=9) | VIT-2763 BID (N=12) | Placebo (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT04364269/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT04364269/SAP_001.pdf